CLINICAL TRIAL: NCT01814891
Title: Determination of Changes in Total Body Stores of Vitamin A in Response to Orange Maize Consumption by Zambian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Zambia II
Record Dates: First submitted 2013-03-07; First posted 2013-03-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Vitamin A Status With Maize Feeding
Keywords: vitamin A; maize; total body reserves; Condition is vitamin A status.; Focus: change in vitamin A status with maize feeding.; Focus: feeding orange maize to children for 90 days.; Focus: total body reserves of vitamin A.
MeSH Terms: conditions — Callosities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Orange maize (Experimental): Children were fed orange maize and the intervention name was "orange"
  Interventions: Other: Orange maize feeding
- Blue vitamin A group (Active Comparator): Received vitamin A in the form of retinyl palmitate in oil at the estimated average requirment.
  Interventions: Other: Vitamin A supplement
- White (Placebo Comparator): Received oil only at the same volume as the vitamin A group
  Interventions: Other: Oil only

INTERVENTIONS:
Other: Orange maize feeding — This group was fed orange maize.
  Arms: Orange maize
Other: Vitamin A supplement — This group received a dose of vitamin A at the estimated average requirement each feeding day of the intervention.
  Arms: Blue vitamin A group
Other: Oil only — This group received a small amount of plain oil without vitamin A.
  Arms: White

SUMMARY:
Determination of liver stores of vitamin A will be determined before and after consumption of high pro-vitamin A orange maize, compared to low provitamin A white maize.

DETAILED DESCRIPTION:
This study will determine the change in total body stores of vitamin A in response to feeding orange maize for 90 days. This will be compared to two other groups of children that are fed white maize, one of which will get a vitamin A supplement at the estimated average requirement.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 57-88 months at the time of initiation of the study
2. Children living in the locality defined by the study and not enrolled in school.
3. Consent from parent/guardian.

Exclusion Criteria:

1. Severely malnourished children (weight for age or height z-scores <-3 standard deviations below the WHO growth reference standards)
2. Children found to be below 57 months and still holding an under five card or above 88 months at the time of initiation of the study or enrolled in school, based on verification of birth dates at screening
3. Children whose families plan to leave the study area before completion of the study
4. Consent not obtained from parent/guardian
5. Children suffering from diarrhea at the time of initiation of the study or with high fever, based on the report of symptoms by the parent/guardian
6. Children with severe anemia (Hb <7.0 g/dL) as determined at the baseline blood draw.

Ages: 57 Months to 88 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Vitamin A status changes | After the intervention, which is approximately 3 months.
  Vitamin A status is measured before and after the intervention.

REFERENCES:
- [Derived] Sheftel J, Valentine AR, Hull AK, Fadjarwati T, Gannon BM, Davis CR, Tanumihardjo SA. Findings in 3 clinical trials challenge the accuracy of the Institute of Medicine's estimated average requirements for vitamin A in children and women. Am J Clin Nutr. 2021 May 8;113(5):1322-1331. doi: 10.1093/ajcn/nqaa132. PMID 32492125
- [Derived] Tanumihardjo SA, Gannon BM, Kaliwile C, Chileshe J, Binkley NC. Restricting vitamin A intake increases bone formation in Zambian children with high liver stores of vitamin. Arch Osteoporos. 2019 Jun 28;14(1):72. doi: 10.1007/s11657-019-0617-y. PMID 31254130
- [Derived] Titcomb TJ, Schmaelzle ST, Nuss ET, Gregory JF 3rd, Tanumihardjo SA. Suboptimal Vitamin B Intakes of Zambian Preschool Children: Evaluation of 24-Hour Dietary Recalls. Food Nutr Bull. 2018 Jun;39(2):281-289. doi: 10.1177/0379572118760373. Epub 2018 Mar 11. PMID 29528727
- [Derived] Suri DJ, Tanumihardjo JP, Gannon BM, Pinkaew S, Kaliwile C, Chileshe J, Tanumihardjo SA. Serum retinol concentrations demonstrate high specificity after correcting for inflammation but questionable sensitivity compared with liver stores calculated from isotope dilution in determining vitamin A deficiency in Thai and Zambian children. Am J Clin Nutr. 2015 Nov;102(5):1259-65. doi: 10.3945/ajcn.115.113050. Epub 2015 Oct 7. PMID 26447158
- [Derived] Mondloch S, Gannon BM, Davis CR, Chileshe J, Kaliwile C, Masi C, Rios-Avila L, Gregory JF 3rd, Tanumihardjo SA. High provitamin A carotenoid serum concentrations, elevated retinyl esters, and saturated retinol-binding protein in Zambian preschool children are consistent with the presence of high liver vitamin A stores. Am J Clin Nutr. 2015 Aug;102(2):497-504. doi: 10.3945/ajcn.115.112383. Epub 2015 Jul 15. PMID 26178727
- [Derived] Gannon B, Kaliwile C, Arscott SA, Schmaelzle S, Chileshe J, Kalungwana N, Mosonda M, Pixley K, Masi C, Tanumihardjo SA. Biofortified orange maize is as efficacious as a vitamin A supplement in Zambian children even in the presence of high liver reserves of vitamin A: a community-based, randomized placebo-controlled trial. Am J Clin Nutr. 2014 Dec;100(6):1541-50. doi: 10.3945/ajcn.114.087379. Epub 2014 Oct 8. PMID 25411289